CLINICAL TRIAL: NCT07041450
Title: A Cohort Study on Screening for Anti-amyloid Treatment Eligibility Using Digital Cognition and Blood-based Biomarkers
Brief Title: Screening for Anti-amyloid Treatment Eligibility Using Digital Cognition and Blood-based Biomarkers
Status: Recruiting | Type: Observational
Sponsor: MoCA Clinic and Institute (Other)
Collaborators: C2N Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: : BBM-01-2025
Record Dates: First submitted 2025-05-07; First posted 2025-06-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Dementia
Keywords: blood-based biomarkers; digital cognitive assessment; diagnostic screening; MoCA; disease-modifying therapy; older adults; early detection; Montreal Cognitive Assessment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants consent for optional storage of 14ml of blood plasma for future biomarker and genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Observational Cohort: The study population will include 500 patients that have been referred to the MoCA Clinic from the Greater Montreal Area. This includes individuals with subjective cognitive decline (SCD), mild cognitive impairment (MCI), and mild dementia.
  Participants complete cognitive tests, health and cognition questionnaires, and undergo a blood test for blood biomarker testing.
  Interventions: Diagnostic Test: Digital MoCA; Diagnostic Test: XpressO; Diagnostic Test: MoCA; Diagnostic Test: Blood-based Biomarkers (BBM); Other: Amyloid Treatment Screening Tool (ATST); Other: MoCA Brain Health Questionnaire (MBHQ); Other: MoCA Medical Questionnaire; Other: Functional Activities Questionnaire+ (FAQ+)
- Paper MoCA Subgroup: Participants will be randomly assigned to complete either the paper MoCA or the digital MoCA Solo at Visit 1, with the other version completed at Visit 2. The Paper MoCA Subgroup will complete the paper MoCA at Visit 1.
  Interventions: Diagnostic Test: Digital MoCA; Diagnostic Test: XpressO; Diagnostic Test: MoCA; Diagnostic Test: Blood-based Biomarkers (BBM); Other: Amyloid Treatment Screening Tool (ATST); Other: MoCA Brain Health Questionnaire (MBHQ); Other: MoCA Medical Questionnaire; Other: Functional Activities Questionnaire+ (FAQ+)
- MoCA Solo Subgroup: Participants will be randomly assigned to complete either the paper MoCA or the digital MoCA Solo at Visit 1, with the other version completed at Visit 2. The MoCA Solo Subgroup will complete the MoCA Solo at Visit 1.
  Interventions: Diagnostic Test: Digital MoCA; Diagnostic Test: XpressO; Diagnostic Test: MoCA; Diagnostic Test: Blood-based Biomarkers (BBM); Other: Amyloid Treatment Screening Tool (ATST); Other: MoCA Brain Health Questionnaire (MBHQ); Other: MoCA Medical Questionnaire; Other: Functional Activities Questionnaire+ (FAQ+)

INTERVENTIONS:
Diagnostic Test: Digital MoCA — A digital version of the Montreal Cognitive Assessment used to evaluate cognitive function. Administered on a tablet at Visit 1 or Visit 2 (randomized).
  Other Names: MoCA Solo
Diagnostic Test: XpressO — A digital cognitive pre-screening tool used to screen for cognitive function. Administered on a tablet at Visit 1.
Diagnostic Test: MoCA — The standard paper-baed Montreal Cognitive Assessment used to evaluate cognitive function. Administered at Visit 1 or Visit 2 (randomized), opposite the digital MoCA.
Diagnostic Test: Blood-based Biomarkers (BBM) — Participants provide a blood sample that is analyzed for Alzheimer's disease-related biomarkers, including PrecivityAD2 and MTBR. These biomarkers are used to assess the biological stage of disease and support diagnostic triage and eligibility assessment for disease-modifying therapy (DMT)
Other: Amyloid Treatment Screening Tool (ATST) — A questionnaire administered to assess eligibility for amyloid-targeted therapies. Both clinician and patient-centered versions are used.
Other: MoCA Brain Health Questionnaire (MBHQ) — A questionnaire designed to capture participants' physical health, emotional well-being, diet, exercise, and social engagement as it relates to cognitive health. Responses are used as part of exploratory analyses to evaluate associations with cognitive status and Alzheimer's disease diagnosis.
Other: MoCA Medical Questionnaire — A structured questionnaire administered to participants to gather information on their medical history, including prior diagnoses, medications, and other health conditions. This data helps to contextualize cognitive symptoms and support diagnostic decision-making in the study.
Other: Functional Activities Questionnaire+ (FAQ+) — A questionnaire designed to assess the participant's ability to perform daily activities, providing insights into their functional status and cognitive impairment. It is a longer version of the original FAQ questionnaire. It is used as part of the screening and exploratory analysis to better understand the relationship between functional abilities and Alzheimer's disease progression.

SUMMARY:
This study evaluates a diagnostic screening solution for Alzheimer's disease (AD) using digital cognitive assessments and blood-based biomarkers. The aim is to reduce time-to-treatment for patients who may benefit from disease-modifying therapy (DMT). The study involves 500 patients referred to the MoCA Clinic in Montreal. Clinical stages will be assessed using digital tools from MoCA Test Inc. (MoCA Cognition), and biological stages via blood biomarkers. Data collected includes demographics, cognitive scores, health questionnaires, biomarker levels, and neurologist-determined eligibility for DMT. The study will result in an algorithm to support diagnostic triage and estimate the efficiency and equity of a fast-track diagnostic pathway. Exploratory endpoints include validation of self-administered digital tools, health-economic estimates, and predictors of cognitive decline.

DETAILED DESCRIPTION:
This study will evaluate a diagnostic screening solution based on clinical and biological stages of Alzheimer's disease (AD) ("Study"). The clinical stages will be screened using the digital tools from MoCA Test Inc. ("MoCA Cognition"). The biological stages will be screened using blood-based biomarkers ("BBM"). Based on the results of this Study, we will establish efficient and equitable criteria for diagnostic triage. The Study will result in an algorithm that can assist in assigning patients into a fast-track diagnostic pathway to determine if they are eligible or not for AD treatment with a disease modifying therapy ("DMT").

Primary objective: To develop and evaluate a diagnostic screening solution based on blood-based biomarkers and digital measures of cognition that could reduce the time-to-treatment for patients who are candidates for AD treatment with a disease modifying therapy.

Primary endpoint: Detailed cohort description of patients referred to the memory clinic MoCA Clinic Inc. ("MoCA Clinic"). This includes: (1) demographic characteristics; (2) cognitive screening scores measured by a digital MoCA via the MoCA score and XpressO application; (3) biomarker levels including PrecivityAD2 and MTBR; (4) the proportion of DMT candidates determined by a neurologist, (5) the causes and frequencies of why patients are not eligible for AD treatment (6) the number of diagnostic follow-up tests required after screening (MRI, PET/CSF), (7) the baseline referral times for future comparison against the fast-track pathway and (8) the time-until-diagnosis.

Secondary endpoints: Based on the primary endpoints, we will estimate the potential benefits of a diagnostic screening solution. This includes an estimation of the number of patients that would potentially miss out on the treatment window in the current diagnostic workflow.

Exploratory endpoints: (1) Validation of a self-administered digital version of the MoCA test ("MoCA Solo") compared to the paper MoCA test, (2) Evaluation of MoCA Solo as digital biomarker within the screening algorithm, (3) Health-economic estimation of the number and costs of follow-up tests at different levels of specificity, (4) The role of age, sex and education on the performance of the screening solution, (5) Prediction of time until patient would progress to moderate dementia based on baseline MoCA score and age, (6) Description of participant's history of symptoms and healthcare usage, (7) Correlation between the patient-centered version and the clinician versions of the Amyloid Treatment Screening Tool (ATST), (8) Evaluate the correlation between the MoCA Brain Health Questionnaire (MBHQ) score and participant diagnosis, (9) Evaluate the effect of the addition of MTBR results into screening algorithm.

Participants: Study population will include 500 patients who have been referred to the MoCA Clinic, including both new patients and existing patients. Based on prior referrals, we anticipate 60% female, 55-90 years, 80% French / 20% English, approximately 20% subjective cognitive decline (SCD), 60% mild cognitive impairment (MCI) and 20% mild dementia.

Study Location: The study is conducted as a single-center study with patients from the Montreal area. Patients will be enrolled at the MoCA Clinic where full informed consent will be obtained.

Study Visits: In the active study period, two MoCA Clinic visits will be planned within 1-3 months: Visit 1 includes data collection feasible at a primary care physician: digital cognitive assessments, blood sample collection and amyloid-treatment screening test. Visit 2 includes cognitive assessment, data collection and diagnosis typical for a neurological visit. After the blood sample is analyzed, the prediction of diagnosis and eligibility for DMT will be made using our algorithm. After the active study period, at 6 months, information from the medical records will be reviewed to evaluate clinical follow-up.

This study is supported by an independent research grant from Eli Lilly Canada Inc.

ELIGIBILITY:
Inclusion Criteria:

* Must be referred to the MoCA Clinic; including both new patients and existing patients who have been seen >1 year ago
* Present with cognitive impairment or cognitive complaints.
* Must have the ability to understand the purpose and risk of the Study and provide informed consent.
* Must have an identified study partner (informant/care partner), who has frequent and sufficient contact with the participant to be able to provide accurate information about the participant's cognitive and functional abilities. The study partner must be available by phone to provide information to the study staff about the participant and agrees to attend one in-person visit at the MoCA Clinic which requires partner input. The study partner should be available for the duration of the study.

Exclusion Criteria:

* An established diagnosis (other than AD), that is a cause for a candidate's cognitive impairment (e.g. substance abuse, cerebrovascular conditions, Lewy body dementia, fronto-temporal dementia, recent head trauma).
* Blood donation (1 unit) within 1 month prior to Study screening.
* Inability to comply with requirements to complete essential components of the Study (e.g. visual impairment, severe kidney disease or ongoing kidney treatment)
* Patients already enrolled in any clinical trial for AD at time of Study screening
* Other unspecified reasons that, in the opinion of the Principal Investigator, or MoCA Clinic and Institute, make the candidate unsuitable for enrolment.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 500 patients that have been referred to the MoCA Clinic from the Greater Montreal Area. There will be a mix of English and French speaking with approximately 80% having French as a first language.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis | From enrollment to 6-month follow-up
  The primary outcome metric is the time to diagnosis for patients that are eligible vs. not eligible for anti-amyloid medication. In this case, time to diagnosis is defined by the time it takes to determine if patient is eligible anti-amyloid medication or not.

SECONDARY OUTCOMES:
Benefit of Diagnostic Screening | Baseline to 6-month follow-up
  This outcome measures the estimated benefit of implementing a diagnostic screening solution by comparing the number of patients who would miss the treatment window for Alzheimer's disease under the current diagnostic workflow versus a hypothetical fast-track workflow incorporating blood-based biomarkers and digital cognitive assessments. The estimate will be based on observed time-to-diagnosis, biomarker results, and predicted disease progression among study participants.

OTHER OUTCOMES:
Validation of MoCA Solo compared to MOCA paper test | Baseline (Visit 1) to 3 months (Visit 2)
  This outcome evaluates the agreement between the self-administered digital MoCA (MoCA Solo) and the traditional paper-based MoCA. The comparison will assess score equivalency, correlation, and potential systematic differences between the two formats to determine if MoCA Solo is a valid alternative for cognitive screening.
Evaluation of MoCA Solo as diagnostic digital biomarker within BBM algorithm | Baseline to 6-month follow-up
  This outcome assesses the utility of the self-administered digital MoCA (MoCA Solo) as a diagnostic digital biomarker when integrated into an algorithm combining cognitive and blood-based biomarker data. Analyses will explore whether MoCA Solo contributes meaningfully to predicting eligibility for disease-modifying therapy (DMT) and staging of Alzheimer's disease.
Accuracy, specificity, and sensitivity of XpressO as compared to the diagnosis of a neurologist. | Baseline
  This outcome evaluates the performance of XpressO, a digital cognitive screening tool and compares it to the findings of a trained neurologist who will identify the clinical stages of Alzheimer's disease. The analysis will help assess the effectiveness of XpressO as a screening tool in the early identification of patients eligible for further cognitive assessment and eventual disease-modifying therapy.
Health-economic estimation of the number and costs of follow-up tests at different levels of sensitivity/specificity for our diagnostic screening solution | Baseline to 6-month follow-up
  This outcome estimates the number and associated costs of follow-up diagnostic tests (e.g., MRI, PET, CSF) that would be required at different levels of sensitivity and specificity of the proposed diagnostic screening solution. The analysis will model how the performance of the screening algorithm impacts healthcare resource use and economic efficiency in the diagnostic workup for Alzheimer's disease.
Impact of Demographics on the Performance of the Diagnostic Screening Algorithm | Baseline to 6-month follow-up
  This outcome evaluates how demographic factors-specifically age, sex, and education level-influence the estimated sensitivity, specificity, and overall performance of the screening algorithm combining cognitive and blood-based biomarkers. The analysis will explore potential differences in diagnostic accuracy across subgroups to assess equity and generalizability of the screening tool.
Prediction of Time to Progression to Moderate Dementia Based on Baseline MoCA Score and Age | Baseline to 6-month follow-up (with predictive modeling beyond observed period)
  This outcome models the expected time until progression to moderate dementia using baseline cognitive performance (MoCA score) and patient age. The analysis will estimate predictive relationships to help identify individuals at higher risk of rapid decline, supporting future applications of the screening algorithm for prognosis and care planning.
Description of Participant Symptom History and Healthcare Utilization | Baseline to 6-month follow-up
  This outcome involves collecting and summarizing participants' self-reported history of cognitive symptoms, duration of concerns, and patterns of healthcare usage related to memory or cognitive issues. Data will include prior visits to healthcare providers, previous diagnostic tests, and timelines from symptom onset to referral, to better understand the diagnostic journey.
Correlation between the patient-centered version and the clinician versions of the Amyloid Treatment Screening Tool (ATST) | Baseline
  This outcome assesses the level of agreement between responses on the patient-centered version and the clinician-administered version of the Amyloid Treatment Screening Tool (ATST). The analysis will evaluate the consistency of reported information and potential discrepancies in determining eligibility for amyloid-targeting therapies.
Correlation between the MoCA Brain Health Questionnaire (MBHQ) score and participant diagnosis | Baseline
  This outcome evaluates the correlation between the MoCA Brain Health Questionnaire (MBHQ) score and the participant's final clinical diagnosis. The analysis will examine how well MBHQ scores align with established diagnostic categories and its potential role as a predictive tool for Alzheimer's disease diagnosis.
Evaluation of the addition of MTBR results into screening algorithm | Baseline to 6-month follow-up
  This outcome evaluates how the inclusion of MTBR (Mitochondrial Tau and Beta-Amyloid Receptor) results improves the diagnostic performance of the screening algorithm. The analysis will assess changes in the algorithm's sensitivity, specificity, and overall accuracy when MTBR biomarkers are integrated, aiming to enhance the early detection of Alzheimer's disease and support better diagnostic triage.

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Nasreddine, MD, Principal Investigator — MoCA Clinic
Locations (1):
- MoCA Clinic and Institute, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Klil-Drori S, Bodenstein KC, Sun S, Kojok L, Gruber J, Ghantous Y, Cummings J, Nasreddine Z. Montreal Cognitive Assessment (MoCA) XpressO: Validation of a digital self-administered cognitive prescreening tool. J Am Geriatr Soc. 2024 Aug;72(8):2516-2522. doi: 10.1111/jgs.18902. Epub 2024 Apr 1. PMID 38558263